CLINICAL TRIAL: NCT06011967
Title: Intubation with Different Angled Intubation Tubes Using C-macr D Blade Videolaringoscope; Evaluation of the Effect on Post-operative Sore Throat, Ease and Time of Intubation, Hoarseness, Subglottic Damage and Hemodynamic Changes : a Prospective Randomized Study
Brief Title: Intubation with Different Angled Intubation Tubes Using C-macr D Blade Videolaringoscope;
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-66175679-514.04.01-788907
Record Dates: First submitted 2023-08-11; First posted 2023-08-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2023-08

CONDITIONS: Intubation; Difficult or Failed; Sore-throat; Hoarseness
Keywords: Videolaryngoscope,; Intubation; C-MAC R Videolaryngoscope,; D- Blade; Subglottic damage; Postoperative sore throat,; Hoarsness
MeSH Terms: conditions — Pharyngitis; Hoarseness

STUDY DESIGN:
Intervention Model Description: In this study we compared the ease of intubation, time needed for intubation, subglottic damage, postoperaitve sore throat, hoarseness and hemodynamic response to orotracheal intubation using three different angled intubation stylets with C-MAC R videolaryngoscope D- blade.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A : 90 degree (Active Comparator): In this group patients were intubated using a 90 degree angled stylet with C-MAC D- Blade videolaryngoscope
  Interventions: Other: Intubation using C-MAC D blade videolariyngoscope
- Group B : 80 degree (Active Comparator): In this group patients were intubated using a 80 degree angled stylet with C-MAC D- Blade videolaryngoscope
  Interventions: Other: Intubation using C-MAC D blade videolariyngoscope
- Group C: 60 degree (Active Comparator): In this group patients were intubated using a 60 degree angled stylet with C-MAC D- Blade videolaryngoscope
  Interventions: Other: Intubation using C-MAC D blade videolariyngoscope

INTERVENTIONS:
Other: Intubation using C-MAC D blade videolariyngoscope — all patients were intubated using the C-MAC D-Blade videolaryngoscope but for each group the intubation tubes were angled in different degrees. First group was intubated using the stylet of 60 degrees, second group was intubated using the stylet of 80 degrees and the third group was intubated using the stylet of 90 degrees.

SUMMARY:
In this study we compared post-operative sore throat, ease and time of intubation, hoarseness, subglottic damage and hemodynamic changes to orotracheal intubation using three different intubation stylets with C-MAC R videolaryngoscope D- blade.

DETAILED DESCRIPTION:
In this study we compared the ease of intubation, time needed for intubation, subglottic damage, postoperaitve sore throat, hoarseness and hemodynamic response to orotracheal intubation using three different intubation stylets with C-MAC R videolaryngoscope D- blade. After the approval of the Ethics Committee, patients were randomized into three groups with closed envelope technique. In Group A endotracheal tube (ETT) is shaped into an angel of 90 degrees, in Group B 80 degrees and in Group C 60 degrees with three different stylets. Laryngoscopy was performed using D-Blade in all 3 groups. Heart rate and blood pressure before and after intubation, time from the entrance of the laryngoscope into the mouth to the passage of the vocal cords, time from the appearance of the cords to intubation, Cormack-Lehane (C-L) classification were recorded. Subglottic damage was examined with fiberoptic bronchoscope. Patients were evaluated regarding postoperative sore throat and hoarsness at 30 minutes, 4, 12, 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA score I-II
* Elective operations
* Supine pozition
* 18-65 years
* No history of surgery in the last 6 months
* No history of airway related surgery
* No anticipated difficult airway

Exclusion Criteria:

* Abdomen, thorax, head-neck surgeries
* Smoker
* Chronic alcohol abuse
* Occupational inhaler agent exposure
* Patients with malignancies
* Patients with a history of radiotheraphy to head-neck region
* Patients with congenital anomalies at head-neck region
* Patients with diagnosed abnormalites of head -neck movements
* Non-cooperatied patients
* Non-oriented patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
sore throat | 30 minutes, 4 hour, 12 hour, 24 hour
  For evaluation of sore throat, the patients were asked whether they had any throat pain. The severity of sore throat was graded as follows: 1: no sore throat, 2: minimal, 3: moderate, 4: severe

SECONDARY OUTCOMES:
Ease of intubation | 2 minutes
  For evaluation of the ease of intubation modified intubation difficulty score was used.
Subglottic damage | 2 hours
  For evaluation of subglottic damage 4-point scaled subglottic damage score was used. grade 0, normal; grade 1, mucosal hyperaemia and oedema and/or slight submucosal haematoma; grade 2, moderately submucosal haematoma; grade 3, mucosal laceration and/or mucosal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Alkım Gizem Yılmaz Selimoğlu, Principal Investigator — Yeditepe University; Ferdi Menda, Prof., Study Director — yYeditepe Universitu
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided